CLINICAL TRIAL: NCT03442205
Title: Randomized Clinical Trial Investigating the Best Method of Treatment of Common Bile Duct Stones
Brief Title: Treatment of Common Bile Duct Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Renyi Qin, Clinical professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJDBPS03
Record Dates: First submitted 2018-02-17; First posted 2018-02-22 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Common Bile Duct Stone
Keywords: Common Bile Duct Stone;; Laparoscopic Common Bile Duct Exploration;; ERCP;
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental)
  Interventions: Procedure: LC + LCBDE + ENBD + primary closure of CBD
- Group B (Experimental)
  Interventions: Procedure: ERCP technique + LC
- Group C (Experimental)
  Interventions: Procedure: LC + LCBDE + primary closure of CBD

INTERVENTIONS:
Procedure: LC + LCBDE + ENBD + primary closure of CBD — LC + LCBDE + ENBD + primary closure of CBD
  Arms: Group A
Procedure: ERCP technique + LC — ERCP technique + LC
  Arms: Group B
Procedure: LC + LCBDE + primary closure of CBD — LC + LCBDE + primary closure of CBD
  Arms: Group C

SUMMARY:
ABSTRACT Introduction: Common bile duct (CBD) stone is a common clinical situation, especially in Asia area. Laparotomy and laparoscopic surgical procedure are often used for treatment. This study compares outcomes of different surgical procedures treating for the disease.

Methods/design: This is a prospective, randomized, controlled multicenter trial with three treatment arms. One group underwent laparoscopic cholecystectomy (LC) + laparoscopic CBD exploration (LCBDE) + intraoperative endoscopic nasobiliary drainage ENBD + primary closure of CBD. The other underwent preoperative endoscopic retrograde cholangiopancreatography (ERCP) and subsequent LC and the third arm underwent laparoscopic cholecystectomy (LC) + laparoscopic CBD exploration (LCBDE) + primary closure of CBD. The duration of the entire trial is two years including prearrangement, follow-up and analyses.

Discussion: Despite the fact plenty evidences provided by meta-analyses suggests that these approaches would appear comparable. It is hopeful to fully address which would be the better approach with this RCT design.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 18 - 80 years.
* Patients diagnosed with gallstones.
* Patients diagnosed with common bile duct stone by one of the three exam (US、MRCP and CT).
* Patients diagnosed with common bile duct stone by intro-operative cholangiography or transcystic exploration.
* Patients understood the trial and accepted one of the three managements.

Exclusion Criteria:

* Combined with Mirizzi syndrome and intrahepatic bile duct stones
* Previous EST/endoscopic retrograde cholangiopancreatography (ERCP) or percutaneous transhepatic biliary drainage (PTBD)
* History of upper abdominal surgery.
* Serious heart, brain, lung, metabolic diseases history.
* Pregnant women.
* Unwillingness or inability to consent for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Adverse outcomes | 24 months
  The patients developing complications/ the total patients

CONTACTS AND LOCATIONS:
Overall Officials: Renyi Qin, pHD, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes